CLINICAL TRIAL: NCT03019939
Title: A Phase II Study of Isavuconazole Prophylaxis in Adult Patients With AML/MDS and Neutropenia
Brief Title: Isavuconazole in Preventing Invasive Fungal Infections in Adult Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome and Neutropenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0373; NCI-2017-00323 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0373 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2021-09-24 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Neutropenia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neutropenia | interventions — isavuconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (isavuconazole) (Experimental): Patients receive isavuconazole PO every 8 hours for 6 doses and then Once a day (QD) or IV over 1 hour every 8 hours for 6 doses and then QD for up to 4 days for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Isavuconazole

INTERVENTIONS:
Drug: Isavuconazole — Given PO or IV
  Other Names: BAL8557

SUMMARY:
This phase II trial studies how well isavuconazole works in preventing invasive fungal infections in adult patients with newly diagnosed acute myeloid leukemia or myelodysplastic syndrome and neutropenia. Isavuconazole may help to prevent invasive fungal infections in adult patients with newly diagnosed acute myeloid leukemia or myelodysplastic syndrome and neutropenia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether prophylaxis with isavuconazole effectively prevents the occurrence of proven or probable invasive fungal infections (IFIs) in patients with newly diagnosed acute myeloid leukemia/myelodysplastic syndrome (AML/MDS) receiving successive cycles of intensive chemotherapy or other therapies for up to 100 days from prophylaxis initiation.

SECONDARY OBJECTIVES:

I. To evaluate the incidence of invasive aspergillosis (IA) within 100 days of beginning isavuconazole prophylaxis in newly diagnosed patients with AML/MDS receiving intensive chemotherapy or other therapies.

II. To evaluate the incidence of other IFIs within 100 days of beginning isavuconazole prophylaxis in newly diagnosed patients with AML/MDS receiving intensive chemotherapy or other therapies.

III. To evaluate the composite outcome of treatment success versus (vs.) failure in this patient population.

IV. To measure the overall survival (OS) of study participants. V. To measure the IFI-free survival of study participants. VI. To document the time to death from any cause in the study population. VII. To document the time to death related to IFI in the study population. VIII. To document the time to diagnosis of proven or probable IFI in the study population.

IX. To document the time to initiation of empiric anti-fungal therapy in the study population.

X. To characterize the safety, tolerability and adverse event (AE) profile of isavuconazole in the prophylactic setting.

EXPLORATORY OBJECTIVES:

I. To assess the potential role, if any, of therapeutic drug monitoring (TDM) of isavuconazole levels in the prophylactic setting in patients with newly diagnosed AML/MDS receiving cytotoxic chemotherapy or other therapies.

II. To determine the in vitro susceptibility of agents causing "breakthrough" IFIs to antifungal agents.

OUTLINE:

Patients receive isavuconazole orally (PO) every 8 hours for 6 doses and then once daily (QD) or intravenously (IV) over 1 hour every 8 hours for 6 doses and then QD for up to 4 days for 12 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either newly diagnosed AML or MDS who have either begun (within 4 days of starting study drug) or are planned to begin specific treatment for their AML/MDS; hydroxyurea and cytarabine used for cytoreduction while awaiting initiation of definitive therapy are not considered "specific" treatment; patients who are participating in other therapeutic clinical trials for their AML/MDS may participate in this trial
* Patients must have or be anticipated to have neutropenia (absolute neutrophil count [ANC] < 0.5 x 10^9/L) (75) for >= 7 days as a result of treatment of their AML/MDS
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Total bilirubin =< 3 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 5 x ULN
* Patients must be able to take oral medications, although a brief period of IV therapy (< 4 days) is permitted at trial entry
* Patients must be willing and able to provide written informed consent for the trial
* Women of childbearing potential (WOCBP) must practice 2 effective methods of birth control during the course of the study; male patients who are partners of WOCBP should also practice an effective method of contraception; effective methods of birth control include diaphragm or condoms with spermicidal foam or jelly, birth control pills (BCPs), injections or patches, intra-uterine devices (IUDs) and surgical sterilization
* Postmenopausal women must be amenorrheic for >= 12 months to be considered of non-childbearing potential
* Women and men must continue birth control for the duration of the trial and >= 3 months after the last dose of study drug
* All WOCBP MUST have a negative pregnancy test prior to first receiving study medication

Exclusion Criteria:

* Proven, probable or possible IFI within the previous 30 days
* Use of any systemic antifungal therapy for > 72 hours during the week prior to study drug initiation
* History of hypersensitivity or idiosyncratic reactions to azoles
* Patients with familial short QT syndrome or with corrected QT (QTc) interval =< 300 ms
* Patients on strong CYP3A4 inducers or inhibitors that cannot be discontinued
* Women who are pregnant or nursing, or intend to be/do so during the course of the study
* Patients with severe hepatic impairment (Child-Pugh class C)
* Patients with known or suspected Gilbert's syndrome at the time of study enrollment
* Patients with known gastrointestinal conditions that could potentially interfere with absorption of orally administered medications
* Any condition that, in the opinion of the investigator, may interfere with the objectives of the study, e.g., any condition requiring the use of prohibited drugs or unstable medical conditions other than AML/MDS, such as a cardiac or neurologic disorder expected to be unstable or progressive during the course of the study (e.g., seizures or demyelinating syndromes, acute myocardial infarction within 3 months of study entry, myocardial ischemia or unstable congestive heart failure, unstable arrhythmias)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prithviraj Bose, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ping Y, Hongmei J, Bellmann C, Ines M, Macmillan T, Webb N, Aram JA, Penack O. A plain language summary on preventing fungal infections with isavuconazole in people with blood-related conditions. Future Microbiol. 2023 Sep;18:861-866. doi: 10.2217/fmb-2022-0280. Epub 2023 Aug 29. PMID 37641932
- [Derived] Bose P, McCue D, Wurster S, Wiederhold NP, Konopleva M, Kadia TM, Borthakur G, Ravandi F, Masarova L, Takahashi K, Estrov Z, Yilmaz M, Daver N, Pemmaraju N, Naqvi K, Rausch CR, Marx KR, Qiao W, Huang X, Bivins CA, Pierce SA, Kantarjian HM, Kontoyiannis DP. Isavuconazole as Primary Antifungal Prophylaxis in Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome: An Open-label, Prospective, Phase 2 Study. Clin Infect Dis. 2021 May 18;72(10):1755-1763. doi: 10.1093/cid/ciaa358. PMID 32236406
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 28, 2017 to July 26, 2019
Groups:
- Prevention (Isavuconazole): Patients receive isavuconazole PO every 8 hours for 6 doses and then QD or IV over 1 hour every 8 hours for 6 doses and then QD for up to 4 days for 12 weeks in the absence of disease progression or unacceptable toxicity.
  Isavuconazole: Given PO or IV
Period: Overall Study
Arm/Group | Prevention (Isavuconazole)
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 34
Age, Continuous [Median (Full Range); unit: years] | 67 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 57
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Proven or Probable Invasive Fungal Infections (IFIs)
Description: Participants with proven or possible invasive fungal infections.
Time Frame: Up to 100 days from prophylaxis initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Participants | 4

2. Secondary Outcome: Number of Participants With Invasive Aspergillosis
Description: Participants with invasive aspergillosissured.
Time Frame: Up to 100 days from prophylaxis initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Participants | 2

3. Secondary Outcome: Number of Participants With Other Invasive Fungal Infections (IFIs)
Description: Participants with other IFIs will be measured.
Time Frame: Up to 100 days from prophylaxis initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Participants | 2

4. Secondary Outcome: Number of Participants With Treatment Success
Description: Will evaluate versus (vs.) failure (defined as Participants with proven or probable IFI, receipt of any other systemic antifungal agent for +/- 4 days for suspected IFI, occurrence of an adverse events possibly or probably related to the study drug resulting in discontinuation of treatment, or withdrawal from the study with no additional follow-up).
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Participants | 46

5. Secondary Outcome: Number of Participants Who Failed Treatment
Description: Will evaluate versus success. Success is defined as Participants with proven or probable IFI, receipt of any other systemic antifungal agent for +/- 4 days for suspected IFI, occurrence of an adverse events possibly or probably related to the study drug resulting in discontinuation of treatment, or withdrawal from the study with no additional follow-up).
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Participants | 19

6. Secondary Outcome: Overall Survival (OS)
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Months | 19.9 [0.9 to 19.9]

7. Secondary Outcome: Invasive Fungal Infections (IFIs)-Free Survival
Description: Time measured in days from start of treatment to IFI or off study date
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Days | 86 [7 to 86]

8. Secondary Outcome: Time to Death From Any Cause
Description: Time to death from any cause will be measured.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Months | 4 [1.1 to 16.4]

9. Secondary Outcome: Number of Participants With Death Related to Invasive Fungal Infections (IFIs)
Description: Death's from invasive fungal infections
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Participants | 0

10. Secondary Outcome: Time to Diagnosis of Proven or Probable Invasive Fungal Infections (IFIs)
Description: Time measured in days from start of treatment to invasive fungal infections
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Days | 24 [7 to 28]

11. Secondary Outcome: Time to Initiation of Empiric Anti-fungal Therapy
Description: Time days from start of empiric anti-fungal therapy.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Prevention (Isavuconazole)
Number analyzed (Participants) | 65
Days | 22 [7 to 80]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Prevention (Isavuconazole)
All-Cause Mortality (participants affected / at risk) | 4/65
Serious Adverse Events (participants affected / at risk) | 30/65
Other Adverse Events (participants affected / at risk) | 14/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Isavuconazole) (N=65)
Abdominal Pain (General disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Death (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 4 (5)
Infection (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 17 (19)
Pain Extremity (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Skin Infection (Infections and infestations) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevention (Isavuconazole) (N=65)
Alanine Aminotransferase Increased (Investigations) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Enlarged Prostate (Reproductive system and breast disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Gastrointestinal Other (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Neutropenic Fever (Blood and lymphatic system disorders) | 7 (8)
Oral Pain (Gastrointestinal disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT03019939/Prot_SAP_000.pdf